CLINICAL TRIAL: NCT06865690
Title: Influence of an Educational Program Utilizing VAK and Kolb's Learning Theories on Basic Cardiopulmonary Resuscitation Knowledge and Practices Among Private Home Nurses in Qatar
Brief Title: Impact of VAK & Kolb-Based Education on CPR Knowledge & Skills Among Private Home Nurses in Qatar
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Collaborators: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Mohamed Elsayed Saad Aboudonya, Resuscitation Training Officer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Qatar; Hamad Medical Corporation (Other: Hamad Medical Corporation)
Record Dates: First submitted 2025-02-14; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: To Evaluate the Impact of a Basic Resuscitation Training Program on the Related Knowledge and Practices of CPR Among Private Home Nurses in Qatar
Keywords: CPR; resuscitation; VAK; KOLB; NURSES; HOME CARE

STUDY DESIGN:
Intervention Model Description: A quasi-experimental (Pre-test and post-test) research design will be utilized in the present study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm Titles: VAK Learning Model Group: Participants receiving CPR training tailored to Fleming's VAK (Experimental): The educational program uses VAK (Visual, Auditory, Kinesthetic) and Kolb's Learning Theories.
- The educational program using VAK (Visual, Auditory, Kinesthetic) and Kolb's Learning Theories. (Experimental): The educational program uses VAK (Visual, Auditory, Kinesthetic) and Kolb's Learning Theories.
  Interventions: Other: Eductional training program

INTERVENTIONS:
Other: Eductional training program — Arms and Interventions
  Arms:
  VAK Learning Model Group:
  Description: Participants in this group will receive an educational program based on Fleming's VAK (Visual, Auditory, Kinesthetic) learning model. The program will tailor teaching methods to participants' sensory preferences (visual, auditory, or kinesthetic).
  Kolb Learning Cycle Group:
  Description: Participants in this group will receive an educational program based on Kolb's Experiential Learning Cycle. The program will emphasize experiential learning through concrete experiences, reflective observation, abstract conceptualization, and active experimentation.
  Interventions:
  VAK Educational Training Program:
  Description: A structured CPR training program designed to align with participants' sensory preferences (visual, auditory, or kinesthetic). The program includes:
  Visual components: Demonstrations, diagrams, and videos.
  Auditory components: Verbal instructions, discussions, and feedback.
  Kinesthetic components: Hands-on
  Arms: The educational program using VAK (Visual, Auditory, Kinesthetic) and Kolb's Learning Theories.

SUMMARY:
Out-of-hospital cardiac arrest (OHCA) is a significant global health challenge, responsible for a substantial proportion of deaths worldwide. Immediate interventions, including cardiopulmonary resuscitation (CPR) and defibrillation, are crucial for achieving optimal outcomes such as restoration of spontaneous circulation (ROSC) and survival until hospital discharge.

Studies reveal that OHCA incidents are prevalent, with an average global incidence rate of 55 cases per 100,000 person-years. In the Gulf Cooperative Council (GCC) region, including Qatar, the majority of OHCA cases occur at home, emphasizing the importance of community-based interventions.

In Qatar, the supreme council of health mandates resuscitation certification for healthcare providers, with renewal periods varying based on the level of the resuscitation.

course. However, private home nurses, who often encounter OHCA cases first, may lack.

adequate CPR training. Unlike Hamad Medical Corporation (HMC) facilities, there are no dedicated CPR trainers for the private healthcare sector.

Training methods incorporating Kolb's Experiential Learning Cycle and Fleming's VAK model can enhance nurses' knowledge and practice. Kolb's model emphasizes experiential learning through reflection and active experimentation, while VAK tailors teaching methods to learners' preferences, including visual, auditory, reading/writing, and kinesthetic styles.

The private healthcare sector in Qatar, with around 5,846 nurses, including approximately 800 providing private nursing services at homes, plays a vital role in delivering healthcare services to the community. However, without adequate CPR training and support, private home nurses may not effectively manage OHCA cases.

To address this gap, it is crucial to establish official CPR training programs for private healthcare sectors, similar to those in HMC facilities. By incorporating diverse learning models and ensuring regular training sessions, private home nurses can acquire the necessary competencies to effectively respond to OHCA incidents, ultimately improving patient outcomes and reducing mortality rates in the community, A quasi-experimental (Pre-test and post-test) research design will be utilized t to evaluate the Influence of VAK and Kolb's Learning Theories on Basic Cardiopulmonary Resuscitation Knowledge and Practices among Private Home Nurses in Qatar. This design facilitates the evaluation of the training's effectiveness by measuring changes in CPR knowledge and skills over time within the same group of nurses. Consequently, it offers valuable insights into the practical outcomes of the training interventions, aligning closely with the study's aim.

DETAILED DESCRIPTION:
1. Introduction/Background Out-of-hospital cardiac arrest (OHCA) is a global health challenge, with an average incidence of 55 cases per 100,000 person-years. In Qatar, OHCA cases are prevalent, with 87.8 per 100,000 population. Most cases occur at home, highlighting the need for community-based CPR training. Private home nurses, who often encounter OHCA cases, lack formal CPR training. This study explores the application of Kolb's Experiential Learning cycle and Fleming's VAK learning model to enhance CPR knowledge and practices among private home nurses in Qatar.
2. Objectives

Primary Objective:

To assess the influence of an educational program on basic CPR knowledge and practices among private home nurses, categorized according to Kolb's Experiential Learning cycle and Fleming's VAK learning model.

Secondary Objectives:

1. Evaluate baseline CPR knowledge and practices before training.
2. Implement and assess the impact of training programs based on Kolb's and VAK models.
3. Compare post-intervention CPR knowledge and practices between the two groups.

3. Study Methodology

Research Design:

A quasi-experimental design with pre-test and post-test assessments will be used. A total of 134 private home nurses will be recruited and divided into two groups:

* Group 1: Trained using Kolb's Experiential Learning Cycle.
* Group 2: Trained using Fleming's VAK learning model.

Data Collection Tools:

1. Tool I: Online questionnaire to assess CPR knowledge, including demographic data, Kolb's LSI, and VAK learning style preferences.
2. Tool II: Observational checklist to evaluate CPR practices (e.g., sequence of steps, quality of chest compressions).
3. Tool III: Observational checklist to assess AED operation skills.

   Training Program:

   - Session 1: Pre-assessment of CPR knowledge and skills (2 hours).
   * Session 2: PowerPoint presentation on CPR and defibrillation (1 hour).
   * Session 3: Hands-on CPR training using ERC's 4-stage approach (3 hours).

   Evaluation :

   Participants will be assessed immediately after training, at 6 months, and at 9 months using the same tools.
4. Study Population and Setting

   Study Population:

   Private home nurses in Qatar are managed by the private nursing sector, Hamad Medical Corporation.

   Inclusion Criteria:
   * Private home nurses with no formal CPR training in the past 12 months.

   Exclusion Criteria:

   - Nurses with formal CPR training in the past 12 months.

   Setting :

   The study will be conducted at the Private Nursing Service building in Medical City, Qatar.
5. Study Procedures

Study Duration:

14 months, including:

* Pre-assessment and piloting: 1 month.
* Training program implementation: 4 months.
* Post-assessments: 4 months (immediate, 6 months, 9 months).
* Data collection and analysis: 4 months.
* Manuscript writing: 2 months.

Informed consent:

Participants will receive detailed information about the study via email and provide voluntary consent before participation.

Confidentiality :

Data will be de-identified, and access will be restricted to the research team.

6. Statistical Analysis Descriptive statistics (e.g., median, frequencies) and inferential statistics (e.g., t-test, Wilcoxon signed-rank test) will be used. Correlation coefficients (Spearman/Pearson) will evaluate relationships between variables. A p-value of ≤0.05 will indicate statistical significance. Data will be analyzed using SPSS software.

7. Ethical Considerations The study will comply with the Declaration of Helsinki, Good Clinical Practice, and Qatar's Ministry of Public Health regulations. Approval will be obtained from the IRB committee at MRC/HMC.

8. Dissemination of Results Findings will be published in scientific journals and presented at conferences. The study is part of a PhD thesis.

ELIGIBILITY:
Inclusion Criteria:

Private home care nurses in Qatar who are interested in participating in the study.

Good knowledge of the English language.

No previous formal CPR training in the past 6 months.

Exclusion Criteria:

Private home care nurses in Qatar who are not interested in participating in the study.

Lack of good knowledge of the English language.

Previous formal CPR training in the past 6 months.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in CPR Knowledge and Practical Skills Score from Baseline to Post-Training at Immediate, 6-Month, and 9-Month Intervals, Assessed by Standardized Questionnaire and Practical Skills Checklist | 9 months
  CPR knowledge will be measured using a standardized multiple-choice questionnaire (MCQ) with a total score range of [0 to 15], and practical skills will be assessed using a CPR skills checklist based on ERC guidelines. Scores greater than 60% will be categorized as satisfactory, and scores less than 60% will be categorized as unsatisfactory. Changes in scores will be measured at three intervals: immediately post-training, at 6 months, and at 9 months.

SECONDARY OUTCOMES:
Baseline CPR Knowledge and Practical Skills Scores of Private Home Nurses | 9 months
  Baseline CPR knowledge will be measured using the standardized MCQ questionnaire, and CPR practical skills will be assessed using the ERC-based skills checklist prior to the educational intervention. Performance will be categorized as satisfactory (>60%) or unsatisfactory (<60%).
CPR Knowledge and Practical Skills Score After Training Based on Kolb's Experiential Learning Cycle at Immediate, 6-Month, and 9-Month Intervals | 9 months
  Post-training CPR knowledge and practical skills will be assessed using the standardized MCQ questionnaire and ERC-based skills checklist among participants trained using Kolb's Experiential Learning Cycle. Performance will be categorized as satisfactory or unsatisfactory at three intervals: immediately post-training, 6 months, and 9 months.
CPR Knowledge and Practical Skills Score After Training Based on Fleming's VAK Learning Model at Immediate, 6-Month, and 9-Month Intervals | 9 months
  Post-training CPR knowledge and practical skills will be assessed using the standardized MCQ questionnaire and ERC-based skills checklist among participants trained using Fleming's VAK learning model. Performance will be categorized as satisfactory or unsatisfactory at three intervals: immediately post-training, 6 months, and 9 months.
Comparison of Post-Training CPR Knowledge and Practical Skills Scores Between Kolb's Experiential Learning Cycle Group and Fleming's VAK Learning Model Group at Immediate, 6-Month, and 9-Month Intervals | 9 months
  The difference in post-training CPR knowledge and practical skills scores between the two groups will be compared using [statistical method, e.g., independent t-test or ANOVA] at three intervals: immediately post-training, 6 months, and 9 months. Performance will be reported as the proportion of participants achieving satisfactory (>60%) or unsatisfactory (<60%) scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP